CLINICAL TRIAL: NCT06313788
Title: Applying a Small Procedure Prior to Injection/Vaccination Reduces Pain Experiences in Child Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lingnan University (Other)
Responsible Party: Principal Investigator, Yeung Wai Lan Victoria, Professor, Lingnan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EC007-2324
Record Dates: First submitted 2024-02-16; First posted 2024-03-15 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Pain
Keywords: mere possession, placebo, analgesia, pain
MeSH Terms: conditions — Agnosia; Pain | interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Masking Description: One group of the participants will be told that they are involved in a marketing survey and will be given a band-aid as a token of appreciation for their participation. This constitutes the mere possession group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Possession Group (Experimental): Participants will be presented with two leaflets about a branded band-aid, which specify its functions, e.g., "stop bleeding", "protect wounds" and "reduce pain". Participants read its analgesic component and mechanism (e.g., "reduces pain sensitization of peripheral nerves") to induce a positive expectation that the branded bandage can effectively help them alleviate pain. Next, participants rate their perceived effectiveness of the band-aid and their use intention. In order to mask the purpose of the study, they will also answer other distractor marketing questions, such as to guess the price of the band-aid and their impression on the package design of the band-aid.
  Participants in possession group will be told that in order to thank them for doing the marketing interview, as a token of appreciation, they will receive a free band-aid with a customized cartoon of their preference.
  Interventions: Other: Possession of a customized placebo analgesic band-aid prior to vaccination or injection
- No Possession Group (No Intervention): Like participants in the possession condition, participants in the no-possession condition will also be first introduced to the function of a branded band-aid using the leaflet advertisement and asked to complete the marketing survey. They will be verbally thanked for their participation to take part in the marketing interview, but they will not be given any first-aid bandage as a souvenir.

INTERVENTIONS:
Other: Possession of a customized placebo analgesic band-aid prior to vaccination or injection — Participants will be told that in order to thank them for doing the marketing interview, as a token of appreciation, they will receive a free band-aid with a customized cartoon of their preference. They will be displayed band-aids with different cartoon images (such as Luffy, minions etc) from which they can freely choose their favorite one . They will be asked to sign their name on the band-aid. This is to establish their sense of ownership. Lastly, with the assistance of the parent, they will be encouraged to anticipate and describe how the owned band-aid is important to them and can help them cope with the forthcoming pain from injection.
  Arms: Possession Group

SUMMARY:
Pain is common among children. Given that children are not as mature and independent in assessing or treating their pain as adults, they are a relatively vulnerable group in terms of pain management and are in need of additional attention. However, there is still insufficient recognition and treatment of pain in children. Taken the procedure of injection/vaccination in children as an example, child patients usually wait for their turn to take the injection from the nurse/doctor, during which anxiety and fear of pain develop. As children are less able to manage their pain than adults, the fear they develop during the waiting time, together with the pain they actually felt after the treatment, can bring negative experiences to them. In this proposed project, the investigators aim to apply a minor procedure prior to a treatment that induces pain (e.g., injection / vaccination) to help managing pediatric pain.

DETAILED DESCRIPTION:
In a series of experiments, Yeung and colleagues found that participants who merely possessed an object framed as having a particular function or benefit experienced an elevation of their self-efficacy in a corresponding domain. For example, participants who possessed reading materials regarded themselves as more knowledgeable. This is because people are inclined to associate themselves with the objects they possess, whose attributes are thus incorporated as part of the self. This mere possession effect also extends to the area of placebo analgesia.

Previous placebo analgesic research typically showed pain reduction after using a placebo analgesic. However, a newly emerged line of research demonstrated that sometimes, people who were merely given possession of a placebo analgesic, without using it, already reported better pain outcomes. This is presumably attributable to the mere possession of the object that enables them to believe they have already received the intended benefit of using it. In Yeung, Geers, and Colloca's study, they found that merely possessing a placebo analgesic yielded placebo analgesia similar to a situation where a placebo analgesic was actually used. The researchers claimed that this observed possession effect was due to the positive expectancy derived from owning a placebo analgesic, i.e., participants expected that the owned placebo analgesic could bring benefits to them.

The finding of the above-mentioned possession-based placebo analgesic effect is encouraging as it can inform healthcare practitioners and physicians about the possibility of tailoring, forming, or optimizing their medical intervention strategies to enhance positive pain outcomes and novel pain management. For instance, practitioners, clinicians, and dentists could consider tailoring their therapeutic interaction and treatment by incorporating an appropriate possession procedure to reduce undesired negative pain outcomes. In this proposed project, the investigators attempt to apply a possession procedure to child patients prior to their treatment that would induce pain.

The investigators hypothesize that acquiring the ownership of a first-aid bandage would contribute to pain alleviation by enhancing children's self-efficacy to cope with pain. The investigators expect that children who receive a first-aid bandage prior to injection would report a lower level of estimated pain (before injection) and lower real-time pain intensity and severity (during injection) than children who do not receive the first-aid bandage prior to the injection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female paediatric patients (aged 6-11 years old) in good general health condition and requiring intramuscular injections
* Submission of signed and dated informed consent form (from paediatric patients and their parents)
* Commitment to comply and cooperate with the implementation of the study procedures

Exclusion Criteria:

* Visual-auditory or neurological deficits
* Allergies to first-aid bandages
* Having existing pain at the injection site

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity Rating (rating how much pain participants feel) | Before injection (5 minutes before injection), during injection (real time) and after injection (1 minute after injection)
  The intensity of pain will be measured by Pain Intensity Numerical Rating Scale (NRS):
  * 5 mins before injection, participants anticipate "how much pain do you expect to have during injection?", using NRS from 0= "No pain at all" to 10= "Extreme pain".
  * During real-time injection, participants report their pain intensity using the same NRS.
  * 1 min after injection: participants report their pain intensity again using the same NRS.
  The higher the NRS rating, the higher the pain intensity.
Pain intensity Measurement (measure how much pain participants feel) | Before injection (5 minutes before injection), during injection (real time) and after injection (1 minute after injection)
  Pain intensity will be measured by the Faces Pain Scale - Revised (FPS-R):
  The scale shows 6 simple cartoon faces, with the face on the far left being expressionless (No pain) and the intensity of pain gradually increasing to the face on the far right showing a very painful expression (Very much pain).
  FPS-R will be used 5 mins before injection, during real-time injection, and 1 min after injection.
  The higher the Visual Analog score, the greater the pain intensity.
Pain Threshold (record the first-time participants feel the pain) | During real time injection, participants will report the first pain sensation they feel (the investigators will record it in milliseconds). It will vary across participants.
  The investigators record the time when the participants first report feeling their initial pain sensation.
  Participants verbally report the point at which they begin to feel pain at the injection site.
  The investigators record the time (in millisecond) participants take to physically perceive a pain sensation from the time of injection.
  The longer/later the time reported means the greater the pain threshold.
Pain unpleasantness (rating how unpleasant participants feel about the pain) | Before injection (5 minutes prior to injection) and after injection (1 minute after injection)
  It measures how emotionally unpleasant participants feel about the pain.
  This is measured by the Visual Analog Scale (VAS): participants draw a cross on a 10 cm line which has a label on the extreme left side stating, "no unpleasant at all", and a label on the extreme right side of the line stating, "the more unpleasant".
  5 mins before injection, participants will estimate their unpleasantness level using the VAS.
  1 min after the injection, participants report their unpleasantness level using the VAS.
  The longer the distance between the far-left point of the line to the cross participants drew, the higher the unpleasantness level.

SECONDARY OUTCOMES:
Mood (rating the positive and negative emotions of the participants) | 1 minute after the manipulation of ownership status
  Participants' positive and negative mood upon obtaining (vs. not obtaining) the ownership of a bandage will be measured by the Positive and Negative Affect Schedule for Children (PANAS-C) Scale
  PANAS-C consists of 9 different descriptors, four of which relates to positive affects, such as "Excited" and the other five relates to negative affects, such as "Upset".
  Participants choose a number that best reflects their current mood for each item (from 1= very slightly or not at all, to 5=extremely).
  The higher the mean score of positive affect items, the more positive emotion the participants feel.
  The higher the mean score of the negative affect items, the more negative emotion the participants feel..
State-anxiety (Rating the participants' current anxiety level) | Baseline, after participants signed the consent form (order is randomized by the computer)
  Participants' state anxiety will be measured by the State-Trait Anxiety Inventory for Children State form (STAIC-S)
  This scale contains 6 statements assessing participants' current state of anxiety. Three items measure the absence of anxiety (e.g., "I feel calm") and the other three items measures the presence of anxiety (e.g., "I feel tense"). Participants use a number from 1 = "Not at all" to 4 = "Very much" to indicate their anxiety level for each item. The absence of anxiety items will be reverse scored.
  The higher the mean rating score, the higher the state anxiety level.
Fear of pain Rating | Baseline, after participants signed the consent form (order is randomized by the computer)
  Participants' fear of pain will be measured by Fear of Pain Questionnaire (FOP).
  FOP contains 30 items describing painful experiences in terms of severe pain, minor pain, medical pain (e.g., "breaking your arm"). Participants rate the extent to which they had a fear of experiencing the pain associated with each item from 1 = "Not at all" to 5 = "Extreme".
  The higher the mean score, the greater the fear of pain.
Magical thinking Rating | Baseline, after participants signed the consent form (order is randomized by the computer)
  Participants' belief that one's ideas, thoughts, actions, words, or use of symbols can influence the course of events in the material world will be measured by the Illusory Beliefs Inventory.
  This scale measures participant's magical thinking including their Magical Beliefs, Spirituality, and Internal State and Thought Action Fusion. It contains 24 items (e.g., "I do something special to prevent bad luck"). Participants rate on a 7-point Likert scale based on their agreement (from 1 = "Strongly disagree" to 7 = "Strongly agree").
  The higher the mean score, the greater the magical thinking tendency.
Pain Self-Efficacy | 1 minute after participants completed the mood scale
  The investigators will use the Pain Self-Efficacy Questionnaire (PSEQ) to measure the confidence level of the participants in handling pain. It contains 8 items. Participants rate how sure they are of being able to do something when they are in pain (from 0= "Not at all confident" to 6=" Completely confident"). For example, "I can cope with my pain without medication."
  The higher the mean score, the greater their perceived self-efficacy in tackling pain.
Self-efficacy to tackle pain | 1 minute after participants completed the Pain Self-Efficacy Questionnaire (PSEQ)
  Participants' self-perceived efficacy concerning their ability to handle the pain will be measured by the Self-Efficacy of Pain Resilience Scale.
  This rating scale measures participants' self-efficacy to handle the pain about injection. For example, "During the injection, I could manage any discomfort". Participants rate on a 7-point Likert scale based on their agreement (from 1= "Strongly disagree" to 7= "Strongly agree").
  The higher the mean score, the greater their perceived self-efficacy in tackling pain.
Expectation of Pain Severity | 5 minutes prior to injection
  Participants will be asked to anticipate "What would be the severity of pain you expect to experience when you receive injection?" from 1 = "No pain at all", to 5 = "Excruciating".
  The higher the score, the greater the expected pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: WAI LAN VICTORIA YEUNG, PhD, Principal Investigator — Lingnan University

IPD SHARING:
Plan to Share IPD: Yes
share all IPD that underlie results in a publication on OSF
Supporting Information: Study Protocol
Time Frame: starting 3 months after publication
Access Criteria: Everyone with access to OSF

REFERENCES:
- [Background] Yeung, V. W. L., Loughnan, S., Kashima, Y., Lun, V. M. C., Yeung, S. S. (2017). When My Object Becomes Me: The Mere Ownership of an Object Elevates Domain Specific Self Efficacy. Applied Psychology, 66(4), 710 741. doi:10.1111/apps.12099
- [Background] Wai-Lan Yeung V, Geers AL, Colloca L. Merely Possessing a Placebo Analgesic Improves Analgesia Similar to Using the Placebo Analgesic. Ann Behav Med. 2020 Sep 1;54(9):637-652. doi: 10.1093/abm/kaaa007. PMID 32227161
- [Background] Yeung, V. W. L., Chan, C. P., Yau, E. K., Lok, W. K., Lun, V. M. C., Chan, E. (2020). I own therefore I can: Efficacy based mere ownership effect. Journal of Experimental Social Psychology, 90, 104005. doi:10.1016/j.jesp.2020.104005
- [Background] Yeung VW, Geers AL. Prior Pain Exposure and Mere Possession of a Placebo Analgesic Predict Placebo Analgesia: Findings From a Randomized, Double-Blinded, Controlled Trial. J Pain. 2021 Apr;22(4):415-431. doi: 10.1016/j.jpain.2020.10.004. Epub 2020 Oct 27. PMID 33127585
- [Background] Yeung VW. Temporal expectancy induced by the mere possession of a placebo analgesic affects placebo analgesia: preliminary findings from a randomized controlled trial. Sci Rep. 2022 Jan 26;12(1):1395. doi: 10.1038/s41598-022-05537-9. PMID 35082351
- [Background] Beggan, J. K. (1992). On the social nature of nonsocial perception: The mere ownership effect. Journal of Personality and Social Psychology, 62(2), 229-237. https://doi.org/10.1037/0022-3514.62.2.229
- [Background] Nesselroade, K. P., Jr., Beggan, J. K., & Allison, S. T. (1999). Possession enhancement in an interpersonal context: An extension of the mere ownership effect. Psychology & Marketing, 16(1), 21-34. https://doi.org/10.1002/(SICI)1520-6793(199901)16:1<21::AID-MAR2>3.0.CO;2-9
- [Background] Laurent, J., Catanzaro, S. J., Joiner, T. E., Jr., Rudolph, K. D., Potter, K. I., Lambert, S., Osborne, L., & Gathright, T. (1999). A measure of positive and negative affect for children: Scale development and preliminary validation. Psychological Assessment, 11(3), 326-338. https://doi.org/10.1037/1040-3590.11.3.326
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Apell, J., Paradi, R., Kokinsky, E., & Nilsson, S. (2011). Measurement of children's anxiety during examination or treatment in hospital--a study evaluating the short-STAI/Matning av barns oro vid undersokning 45 eller behandling pa sjukhus--en studie som utvarderar short STAI. Nursing Science & Research in the Nordic Countries, 31(1), 45+. https://link.gale.com/apps/doc/A273786636/HRCA?u=anon~691011a5&sid=googleScholar&xid=05fcdcaa
- [Background] Vambheim SM, Lyby PS, Aslaksen PM, Flaten MA, Asli O, Martinussen LM. The Fear of Pain Questionnaire-III and the Fear of Pain Questionnaire-Short Form: a confirmatory factor analysis. J Pain Res. 2017 Aug 8;10:1871-1878. doi: 10.2147/JPR.S133032. eCollection 2017. PMID 28860842
- [Background] Kingdon BL, Egan SJ, Rees CS. The Illusory Beliefs Inventory: a new measure of magical thinking and its relationship with obsessive compulsive disorder. Behav Cogn Psychother. 2012 Jan;40(1):39-53. doi: 10.1017/S1352465811000245. Epub 2011 May 16. PMID 21729346
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Hanssen MM, Peters ML, Vlaeyen JWS, Meevissen YMC, Vancleef LMG. Optimism lowers pain: evidence of the causal status and underlying mechanisms. Pain. 2013 Jan;154(1):53-58. doi: 10.1016/j.pain.2012.08.006. Epub 2012 Oct 18. PMID 23084002